CLINICAL TRIAL: NCT03731260
Title: A 3-Part, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate Safety and Efficacy of Avapritinib (BLU-285), a Selective KIT Mutation-Targeted Tyrosine Kinase Inhibitor, in Indolent and Smoldering Systemic Mastocytosis With Symptoms Inadequately Controlled With Standard Therapy
Brief Title: (PIONEER) Study to Evaluate Efficacy and Safety of Avapritinib (BLU-285), A Selective KIT Mutation-targeted Tyrosine Kinase Inhibitor, Versus Placebo in Patients With Indolent Systemic Mastocytosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLU-285-2203; 2018-000588-99 (EudraCT Number)
Record Dates: First submitted 2018-10-30; First posted 2018-11-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Indolent Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic | interventions — avapritinib

STUDY DESIGN:
Intervention Model Description: In Part 1 of the study, patients will be randomly assigned to 1 of 3 doses of avapritinib or to placebo + BSC. Once the recommended phase 2 dose (RP2D) of avapritinib is identified in Part 1, patients in Part 2 will be randomly assigned to receive avapritinib at the RP2D + BSC or matching placebo + BSC. In Part 3, patients who have completed treatment in Part 1 or Part 2 of the study (including those initially randomized to placebo) may participate in a long-term open-label extension, receiving avapritinib at the RP2D + BSC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- (Part 1) Avapritinib Dose 1 + BSC (Experimental): Avapritinib will be administered orally in continuous 28-day cycles
  Interventions: Drug: Avapritinib
- (Part 1) Avapritinib Dose 2 + BSC (Experimental): Avapritinib will be administered orally in continuous 28-day cycles
  Interventions: Drug: Avapritinib
- (Part 1) Avapritinib Dose 3 + BSC (Experimental): Avapritinib will be administered orally in continuous 28-day cycles
  Interventions: Drug: Avapritinib
- (Part 1) Placebo + BSC (Placebo Comparator): Placebo will be administered orally in continuous 28-day cycles
  Interventions: Drug: Placebo
- (Part 2) Avapritinib RP2D + BSC (Experimental): Avapritinib will be administered orally in continuous 28-day cycles
  Interventions: Drug: Avapritinib
- (Part 2) Placebo + BSC (Placebo Comparator): Placebo will be administered orally in continuous 28-day cycles
  Interventions: Drug: Placebo
- (Part 3) Avapritinib RP2D + BSC (Experimental): Avapritinib will be administered orally in continuous 28-day cycles
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — Avapritinib tablet
  Other Names: BLU-285
  Arms: (Part 1) Avapritinib Dose 1 + BSC; (Part 1) Avapritinib Dose 2 + BSC; (Part 1) Avapritinib Dose 3 + BSC; (Part 2) Avapritinib RP2D + BSC; (Part 3) Avapritinib RP2D + BSC
Drug: Placebo — Placebo tablet
  Arms: (Part 1) Placebo + BSC; (Part 2) Placebo + BSC

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study comparing the efficacy and safety of avapritinib + best supportive care (BSC) with placebo + BSC in patients with indolent systemic mastocytosis (ISM) whose symptoms are not adequately controlled by BSC. The study will be conducted in 3 parts. All patients will receive treatment with avapritinib during Part 3 including those rolling over from the placebo group.

ELIGIBILITY:
Key Inclusion Criteria:

* 1. Patient must have SM, confirmed by Central Pathology Review of BM biopsy, and central review of B- and C-findings by WHO diagnostic criteria.
* 2. Patient must have moderate-to-severe symptoms based on minimum mean total symptom score (TSS) of the ISM Symptom Assessment Form (ISM-SAF) over the 14-day eligibility screening period.
* 3. Patient must have failed to achieve adequate symptom control for 1 or more Baseline symptoms.
* 4. For patients receiving corticosteroids, the dose must be ≤ 20 mg/d prednisone or equivalent, and the dose must be stable for ≥ 14 days.
* 5. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.

Key Exclusion Criteria:

* 1. Patient has been diagnosed with any of the following WHO SM subclassifications: cutaneous mastocytosis only, smoldering SM, SM with associated hematologic neoplasm, aggressive SM, mast cell leukemia, or mast cell sarcoma.
* 2. Patient must not have received prior treatment with avapritinib.
* 3. Patient must not have had any cytoreductive therapy including but not limited to masitinib and midostaurin, or investigational agent for < 14 days or 5 half-lives of the drug (whichever is longer), and for cladribine, interferon alpha, pegylated interferon, or antibody therapy < 28 days or 5 half-lives of the drug (whichever is longer), before beginning the 14-day ISM-SAF eligibility TSS assessment.
* 4. Patient must not have received radiotherapy or psoralen and ultraviolet A (PUVA) therapy < 14 days before beginning the 14-day ISM-SAF eligibility TSS assessment.
* 5. Patient must not have received any hematopoietic growth factor the preceding 14 days before beginning the 14-day ISM-SAF eligibility TSS assessment.
* 6. Patient must not have a QT interval corrected using Fridericia's formula (QTcF) of > 480 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Part 1: Recommended Phase 2 dose (RP2D) in patients with ISM | 9 months
Part 2: Mean change in ISM Symptom Assessment Form (ISM-SAF) total symptom score (TSS) as compared to placebo | 6 months
  0 - 110 points (higher value represents worse symptom outcomes)
Part 3: Number of Participants with Adverse Events | Up to 5 years

SECONDARY OUTCOMES:
Part 2: Proportion of patients with a ≥50% reduction in serum tryptase | 6 months
Part 2: Proportion of patients with a ≥50% reduction in peripheral blood V-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog aspartate 816 valine (KIT D816V) allele fraction or undetectable for patients with detectable mutation at Baseline | 6 months
Part 2: Proportion of patients with ≥50% reduction in ISM-SAF TSS | 6 months
Part 2: Proportion of patients with ≥30% reduction in ISM-SAF TSS | 6 months
Part 2: Proportion of patients with a ≥50% reduction in bone marrow mast cells or no aggregates for patients with aggregates at Baseline | 6 months
Parts 1, 2, and 3: Change in serum tryptase | Up to 5 years
Parts 1, 2, and 3: Change in KIT D816V allele burden in blood | Up to 5 years
Parts 1, 2, and 3: Change in bone marrow mast cells | Up to 5 years
Parts 1, 2, and 3: Change in best supportive care (BSC) concomitant medication usage | Up to 5 years
Parts 1, 2, and 3: Change from Baseline in ISM-SAF Score | Up to 5 years
Parts 1, 2, and 3: Change in Mastocytosis Quality of Life Questionnaire (MC-QoL) | Up to 5 years
Parts 1, 2, and 3: Change in Patient's Global Impression of Symptom Severity (PGIS) | Up to 5 years
Parts 1, 2, and 3: Change in 12-item Short Form Health Survey (SF-12) | Up to 5 years
  0 - 100 points (higher value represents better symptom outcomes)
Parts 1, 2, and 3: Change in Patients' Global Impression of Change (PGIC) | Up to 5 years
  1 - 7 (higher value represents worse symptom outcomes)
Parts 1, 2, and 3: Change in EuroQuol 5 Dimensions 5 Levels (EQ 5D-5L) | Up to 5 years
  0 - 100 (higher value represents better symptom outcomes)
Parts 1, 2, and 3: Safety of avapritinib as assessed by number of adverse events | Up to 5 years
  CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (49):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Stanford Cancer Institute, Stanford, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Michigan Medicine, University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Health System (DUHS), Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- University Hospital Antwerp, Edegem, Belgium
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Michael's Hospital, Toronto, Ontario
- Odense Universitetshospital, ORCA/Allergicentret, Hudafdeling I og Allergicenter, Odense, Denmark
- France (3):
  - Hôpital de la Timone, Service de dermatologie, Marseille
  - Hôpital Pitié-Salpêtrière, Service de Dermatologie, Paris
  - CHU Toulouse Larrey, CEREMAST, Service de Dermatologie et Allergologie cutanée, Toulouse
- Germany (7):
  - Uniklinik RWTH Aachen, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - University Clinic Hamburg Eppendorf, University Cancer Center Hamburg (UCCH), Hamburg
  - Universitätsklinikum Schleswig-Holstein, Hämatologie/Onkologie, Lübeck
  - Universitätsklinik Mainz, Universitäts-Hautklinik, Clinical Research Center, Mainz
  - Universitätsmedizin Mannheim, III. Medizinische Klinik, Mannheim
  - Klinikum rechts der Isar, Technische Universität München, Munich
- Italy (4):
  - A.O.U di Bologna - IRCCS, Istituto di Ematologia Lorenzo e Ariosto Seragnoli, Ematologia, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Poloclinico, UOC Ematologia, Milan
  - A.O. OO.RR. S.Giovanni di Dio e Ruggi d'Aragona, University of Salerno, Salerno
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Netherlands (2):
  - University Medical Center Groningen (UMCG), Groningen
  - Erasmus Medical Center, Rotterdam
- Oslo Universitetssykehus, Rikshospitalet, Department of Hematology, Oslo, Norway
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - lnstituto de Estudios de Mastocitosis de Castilla la Mancha, Hospital Virgen del Valle - Complejo Hospitalario de Toledo, Toledo
- Sweden (2):
  - Karolinska University Hospital, Hematologimottagningen R51, Stockholm
  - Akademiska sjukhuset, Hematologmottagningen/101A, Uppsala
- University Hospital Basel, Basel, Switzerland
- United Kingdom (3):
  - NHS Greater Glasgow and Clyde, Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral

REFERENCES:
- [Derived] Worth S, George TI, Shaheen DJ, Roche M, Vachhani P. Chronic Anaphylaxis With Indolent Systemic Mastocytosis: A Case Report. Case Rep Hematol. 2025 Nov 6;2025:9562195. doi: 10.1155/crh/9562195. eCollection 2025. PMID 41244098
- [Derived] Gotlib J, Castells M, Elberink HO, Siebenhaar F, Hartmann K, Broesby-Olsen S, George TI, Panse J, Alvarez-Twose I, Radia DH, Tashi T, Bulai Livideanu C, Sabato V, Heaney M, Van Daele P, Cerquozzi S, Dybedal I, Reiter A, Pongdee T, Barete S, Ustun C, Schwartz L, Ward BR, Schafhausen P, Vadas P, Bose P, DeAngelo DJ, Rein L, Vachhani P, Triggiani M, Bonadonna P, Rafferty M, Butt NM, Oh ST, Wortmann F, Ungerstedt J, Guilarte M, Taparia M, Kuykendall AT, Arana Yi C, Ogbogu P, Gaudy-Marqueste C, Mattsson M, Shomali W, Giannetti MP, Bidollari I, Lin HM, Sulllivan E, Mar B, Scherber R, Roche M, Akin C, Maurer M. Avapritinib versus Placebo in Indolent Systemic Mastocytosis. NEJM Evid. 2023 Jun;2(6):EVIDoa2200339. doi: 10.1056/EVIDoa2200339. Epub 2023 May 23. PMID 38320129
- [Derived] Padilla B, Shields AL, Taylor F, Li X, Mcdonald J, Green T, Boral AL, Lin HM, Akin C, Siebenhaar F, Mar B. Psychometric evaluation of the Indolent Systemic Mastocytosis Symptom Assessment Form (ISM-SAF) in a phase 2 clinical study. Orphanet J Rare Dis. 2021 Oct 18;16(1):434. doi: 10.1186/s13023-021-02037-3. PMID 34663404